# STATISTICAL ANALYSIS PLAN

# LA55-0417

Safety and efficacy of early-start deferiprone treatment in infants and young children newly diagnosed with transfusion-dependent beta thalassemia

Final Version 1

24 SEP 2020

# Approved by

David Lee, Ph.D.

Scientific Leader, Biostatistics

Chiesi Canada Corp.

24 SÆP 2020

Date (DD MMM YYYY)

Anna Rozova, MD Director, Medical Safety

Chiesi Canada Corp.

Date (DD MMM YYYY)

Fernando Tricta, MD

Senior Vice President, Medical Affairs

Chiesi Canada Corp.

Date (DD MMM YYYY)

# **Table of Contents**

| | Title | e page | | 1 |
|---|---|---|---|---|
| | App | rovals | | 2 |
| | List | of Abbi | reviations | 5 |
| 1. | | | n | |
| 2. | Stud | ly Obje | ctives | 8 |
| | 2.1 | Prima | ry Objective | 8 |
| | 2.2 | | dary Objective | |
| 3. | Stud | | n | |
| | 3.1 | - | ption of Study Design | |
| | 3.2 | | per of Patients. | |
| | 3.3 | | Procedures | |
| 4. | | • | nts and Evaluations | |
| | 4.1 | | cy Measurements | |
| | | 4.1.1 | Serum Ferritin (µg/L) | |
| | | 4.1.2 | Transferrin Saturation (%) | |
| | | 4.1.3 | Labile Plasma Iron (µM) | 15 |
| | 4.2 | Safety | Measurements | 16 |
| | | 4.2.1 | Medical Events, Adverse Events, and Serious Adverse Events | 16 |
| | | 4.2.2 | Laboratory Measurements | 16 |
| | | 4.2.3 | Physical Examinations | 17 |
| | | 4.2.4 | Vital Signs | 17 |
| | | 4.2.5 | Concomitant Medications | 17 |
| <b>5.</b> | Stat | istical A | analysis | 18 |
| | <b>5.1</b> | Study | Populations | 18 |
| | | 5.1.1 | Intent-to-Treat Population | 18 |
| | | 5.1.2 | Per Protocol Population | 18 |
| | | 5.1.3 | Safety Population | 18 |
| | <b>5.2</b> | Effica | cy Endpoints | 18 |
| | | 5.2.1 | Primary Efficacy Endpoint | 18 |
| | | 5.2.2 | Secondary Efficacy Endpoints | 19 |

| 5.3 | Safety | 19 | |
|------|--------|-------------------------------------------------|-------|
| 5.4 | Patier | nt Disposition and Drug Exposure | 19 |
| 5.5 | Patier | 19 | |
| 5.6 | Analy | 20 | |
| 5.7 | Analy | 22 | |
| | 5.7.1 | AEs and SAEs | 22 |
| | 5.7.2 | Number of discontinuations due to AEs | |
| | 5.7.3 | Hematology and biochemistry | 23 |
| | 5.7.4 | Urinalysis | 23 |
| | 5.7.5 | Vital signs | 23 |
| | 5.7.6 | Prior and concomitant medications | 24 |
| | 5.7.7 | Time to withdrawal | 24 |
| | 5.7.8 | Height and weight | |
| SUMM | IARY T | ABLES AND FIGURES | 25 |
| 14.1 | Patier | nt disposition, demographics, and baseline data | 25 |
| 14.2 | Effica | ıcy analyses | 25 |
| 14.2 | 2.1 | Serum ferritin (µg/L) | 25 |
| 14.2 | 2.2 | Labile plasma iron (µM) | |
| 14.2 | 2.3 | Transferrin saturation (%) | |
| 14.3 | Safety | y analyses | 26 |
| 14.3 | _ | Adverse events | |
| 14.3 | 3.2 | Vital signs | 27 |
| 14.3 | 3.3 | Height | |
| 14.3 | 3.4 | Weight | |
| 14.3 | 3.5 | Concomitant medications | |
| 14.3 | 3.6 | Laboratory data | 28 |
| | 14.3.6 | 5.1 Hematology | |
| | | 5.2 Biochemistry | |
| 14.3 | | Prolactin | |
| 14.4 | Other | analyses | 28 |
| 14.2 | | ıcy | |
| 14.3 | | y | |
| | ~ arti | <del>,</del> | ····· |

| 14.3.1 | Hematology | 29 |
|------------|--------------------------------------------------|----|
| 14.3.2 | Biochemistry | 29 |
| DATA LISTI | NGS | 30 |
| TABLE SHE | LLS | 32 |
| 14.1 Pati | ent disposition, demographics, and baseline data | 33 |
| 14.2 Effic | cacy Analyses | 39 |
| 14.2.1 | Serum Ferritin (µg/L) | 39 |
| 14.2.2 | Labile Plasma Iron (μM) | |
| 14.2.3 | Transferrin Saturation (%) | 47 |
| 14.3 Safe | ty analyses | 51 |
| 14.3.1 | Adverse events | 51 |
| 14.3.2 | Vital signs | 54 |
| 14.3.3 | Height | 56 |
| 14.3.4 | Weight | 59 |
| 14.3.5 | Concomitant medications | 62 |
| 14.3.6 | Laboratory data | 63 |
| 14.3 | .6.1 Hematology | 63 |
| | .6.2 Biochemistry | |
| 14.3.7 | Prolactin | 70 |
| 14.4 Oth | er analyses | 71 |

# **List of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| ADR | adverse drug reaction |
| AE | adverse event |
| ALT | alanine transaminase |
| ANC | absolute neutrophil count |
| ANCOVA | analysis of covariance |
| AST | aspartate transaminase |
| CS | clinically significant |
| CI | confidence interval |
| CRA | clinical research associate |
| CRF | case report form |
| CRO | contract research organization |
| CRP | C-reactive protein |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transpeptidase |
| HIV | human immunodeficiency virus |
| HPLC | high performance liquid chromatography |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ITT | intent-to-treat |
| LPI | labile plasma iron |
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCS | not clinically significant |
| NTBI | non-transferrin-bound iron |
| PP | per protocol |
| PT | preferred term |
| RBC | red blood cell |
| SADR | serious adverse drug reaction |

# Chiesi Canada Corp.

| Abbreviation | Definition |
|--------------|---------------------------|
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SF | serum ferritin |
| SOC | system organ class |
| t.i.d | three times a day |
| TSAT | transferrin saturation |
| ULN | upper limit normal |
| WBC | white blood cell |
| WHO | World Health Organization |

#### 1. Introduction

This document outlines the statistical analysis plan (SAP) for clinical study LA55-0417, titled "Safety and efficacy of early-start deferiprone treatment in infants and young children newly diagnosed with transfusion-dependent beta thalassemia".

The SAP details the statistical methods to be used in analyzing the data from the study, and presents the mock-up tables that will be included in the clinical study report. When the SAP and the clinical study protocol are different with respect to the planned analyses, the SAP is to supersede the clinical study protocol.

The standards used to compile the clinical data will be based on the Study Data Tabulation Model v1.4, SDTM implementation guide v 3.2 as well as controlled terminology v 2017-06-30 from the Clinical Data Interchange Standards Consortium (CDISC). Tables, listings and figures will be programmed using data from the SDTM datasets.

# 2. Study Objectives

### 2.1 Primary Objective

To evaluate the effect of early treatment with deferiprone on lessening progressive iron overload in infants and young children with transfusion-dependent  $\beta$ -thalassemia.

# 2.2 Secondary Objective

To evaluate the safety and tolerability of early treatment with deferiprone in infants and young children with transfusion-dependent  $\beta$ -thalassemia.

# 3. Study Design

### 3.1 Description of Study Design

This is a multi-center, randomized, double-blind, placebo-controlled study in infants and young children newly diagnosed with transfusion-dependent  $\beta$ -thalassemia. Patients start on a red blood cell (RBC) transfusion regimen designed to maintain a hemoglobin level > 9 g/dL, but still have a serum ferritin level well below the threshold that current treatment guidelines state should be reached before iron chelation therapy can begin.

Screening is conducted within 14 days prior to the start of dosing. At baseline, eligible participants are randomized in a 1:1 ratio to receive either deferiprone oral solution 80 mg/mL or matching placebo. Visits are scheduled approximately monthly (every 30 ±10 days) for the determination of levels of serum ferritin (SF), labile plasma iron (LPI), and transferrin saturation (TSAT), and for assessments of safety that include determination of liver enzymes (ALT and AST) and growth measurements.

Dosage begins at 25 mg/kg/day, divided into 3 doses (t.i.d.), and is increased to 50 mg/kg/day (divided t.i.d.) after 2 weeks. After that, it is increased to 75 mg/kg/day (divided t.i.d.) for patients who meet either of the following criteria:

- An SF value  $\geq 800 \,\mu\text{g/L}$  (but still below 1000  $\,\mu\text{g/L}$ ) and/or an LPI value  $\geq 0.6 \,\mu\text{M}$  and/or a TSAT value  $\geq 60\%$  at 2 consecutive visits, or
- An increasing trend in any of the above 3 measures (SF, LPI, and/or TSAT) at 3 consecutive visits, regardless of value

If a single occurrence of any of the following is detected at any time, treatment is interrupted:

- SF value below the lower reference range for the child's age
- Mild neutropenia, defined as an absolute neutrophil count (ANC)  $< 1.5 \times 10^9$ /L but  $> 1.0 \times 10^9$ /L
- Fever or other signs of infection, prior to confirmation that ANC is  $\geq 1.5 \times 10^9/L$

As these parameters are known to fluctuate, the assessment is repeated as soon as possible to verify that treatment interruption is necessary. Treatment is re-initiated after the abnormally low SF or ANC level is recovered, or when the fever or infection resolves or is determined to not be indicative of neutropenia.

If moderate neutropenia (ANC  $\leq 1.0 \times 10^9/L$ ) is confirmed, the patient is withdrawn from the study.

Patients remain in the study for 12 months or until their SF level is found to be  $\geq$  1000 µg/L at 2 consecutive visits, whichever comes first. Since SF level may be impacted by the presence of infection, it must additionally be verified that the child has had no signs of infection in the previous 7 days, including the day of the visit, and that the level of C-reactive protein (CRP) is no greater than 20% higher than the normal range for the patient's age. If there are signs of infection and/or the CRP level is above this threshold, the SF level must be checked again a minimum of one week later. (**Note:** If an investigator has valid reason to believe that an SF level  $\geq$  1000 µg/L may be attributable to infection even if this is not indicated by the CRP result, SF may be rechecked once more a minimum of one week later.)

#### 3.2 Number of Patients

A planned total of 64 patients are to be enrolled in the study, 32 in each arm.

# 3.3 Study Procedures

The procedures and assessments to be conducted at each study visit are shown in Table 1.

# Remote patient visits due to the COVID-19

Due to the COVID-19 pandemic, some patients were unable to attend the site due to transportation disruptions, site restrictions/availability and to maintain social distancing. In cases where patients are unable to attend the site due to COVID-19 restrictions, remote patient visits have been performed as follows:

- Patients were contacted and verbally consented to having their visits performed remotely, including having lab samples collected from Al Mokhtabar /Prodia phlebotomists at their home (if Al Mokhtabar /Prodia cannot continue at home visits, the patients will have to attend the closest local branch), and IP delivered, and completed patient diary cards and used/unused IP from the last visit collected by the courier. This discussion occurred before any aspect of remote visits occurred and was documented in the source
- The patient was called by the PI/delegated site staff for their remote visit. These calls must be documented in the source.
- Recommendation that the site try to use the later dates within the visit windows to have visits.
- Sample collection: weekly, bi-weekly and monthly samples (CBCs, biochemistry, LPI, serum ferritin, C-reactive protein, transferrin saturation and CRP if applicable) were collected by AM/Prodia phlebotomists at the patients' homes and/or local branch.

### It is noted that:

- The morning dose should be taken AFTER these samples are collected. Therefore, the samples should have been collected in the morning.
- Review of the results within 24 hours of receipt is still in effect.
- If a transfusion was scheduled on the day of the visit, the blood samples for serum ferritin, LPI, and TSAT must have been collected before the transfusion was performed.
- Dose escalations and withdrawal criteria remained unchanged.
- LPI samples were collected in both Indonesia and Egypt as per protocol, however, shipments were suspended due to Covid-19 and the third-party analysis laboratory, Radbound, had closed until 28 APR 2020.
- PI/site staff reviewed and followed up on: Transfusion history, AE/SAEs and concomitant medication, exposure and dosing.
- All study reminders were communicated to the patients.
- If possible M12 and/or Early Termination Visits (within 30 days of the last dose) were conducted on-site. These have more time sensitive collections for prolactin.
- If possible, patients were asked to perform the following assessments and share the information over the phone during the visit: Patient's body temperature taken with the thermometers provided at study start; Measurement height/length: using string and/or tape measure.

IP and patient diary card:

- IP was called from IVRS by the site staff using the weight from the last on-site visit.
- Only a 1-month supply was provided to the patient as per protocol.
- IP accountability was maintained via the logs as per usual.
- IP and blank patient diary card were collected by courier arranged by EPx/Sydna and transported to the patients' home:
- The patients: verbally consented to allowing IP to be delivered, understanding that their address will be shared with the courier; and that they must sign for the IP upon receipt.
- The courier used temperature monitoring devices (TMD), which were stopped when IP is delivered.
- The patients did not begin the new medication until the TMD readings were downloaded and verified by Chiesi Canada Corp.
- The site printed off the IVRS report for IP dispensation and wrote the TMD used for each shipment. This is to be filed in the patient binder.
- Used and unused IP and the patient diary card from the previous visit were returned
  to the site via courier. The site reviewed the compliance and patient diary card for
  AEs/SAEs, concomitant medications and exposure and contacted the patient if
  needed to clarify any information recorded.

The sites must clearly document which patients were participating in remote visits, and which assessments were not collected as per protocol. Potential protocol deviations following the above process must be documented and can include heart rate and blood pressure not collected, physical exam not performed, visits out of window due to Covid-19 and weight (weight from the previous on-site visit to be used for dispensation/dosing if unable to be collected during remote visit).

Once Covid-19 restrictions are lifted, on-site study visits are to resume.

 Table 1
 Table of study procedures

| | Day -14<br>to 0<br>(Screenin<br>g) | Day 0 | Month<br>1 1 | Month 2 | Month 3 | Month<br>4 | Mont<br>h 5 | Month<br>6 | Month<br>7 | Month<br>8 | Month<br>9 | Month<br>10 | Month<br>11 | Month 12 or End of Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent/<br>assent | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Eligibility criteria | X | V | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | |
| Hematology <sup>3</sup> | X | X | Weekl | y (±3 days | s) after sta | art of dosi | ng up to N | Month 6 | Biwee | kly (±3 da | ys) until t | erminatio | n from th | e study |
| Blood chemistry 4,5 | X | | X | | X | | | X | | | X | | | X |
| DNA testing (if applicable) <sup>6</sup> | X | | | | | | | | | | | | | |
| Urinalysis 5,7 | X | | | | | | | | | | | | | X |
| Serology <sup>8</sup> | X | | | | | | | | | | | | | |
| Physical examination <sup>5</sup> | X | | X | | X | | | X | | | X | | | X |
| Vital signs <sup>9</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height <sup>10</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Labile plasma iron | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | Day -14<br>to 0<br>(Screenin<br>g) | Month<br>0,<br>Day 0<br>(Baselin<br>e) | Month<br>1 1 | Month 2 | Month<br>3 | Month<br>4 | Mont<br>h 5 | Month<br>6 | Month<br>7 | Month<br>8 | Month<br>9 | Month<br>10 | Month<br>11 | Month 12 or End of Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Transferrin saturation 11 | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum ferritin <sup>11</sup> Prolactin <sup>12</sup> | X | X<br>X | X | X | X | X | X | X | X | X | X | X | X | X<br>X |
| Dispense study medication | | X | X | X | X | X | X | X | X | X | X | X | X | |
| Provide diary card | | X | X | X | X | X | X | X | X | X | X | X | X | |
| Dosing 13 | | | | | Three t | imes daily | from bas | eline until | terminat | ion from t | he study | <u> </u> | | |
| Review and collect diary card | | | X | X | X | X | X | X | X | X | X | X | X | X |
| Collect study<br>medication<br>containers | | | X | X | X | X | X | X | X | X | X | X | X | X |
| Assess treatment compliance | | | X | X | X | X | X | X | X | X | X | X | X | X |
| Prior & concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Medical events | X | X | | | | | | | | | | | | |
| Adverse events | Throughout the study after start of dosing | | | | • | • | | | | | | | | |
| Transfusion<br>history | | • | | | | Γ | Throughou | it the stud | y | | | | | |

#### V: Verify

- Visits are scheduled every 30 days ( $\pm$  10 days).
- Patients terminate from the study at Month 12 or when they have been found to have a serum ferritin level  $\geq$  1000  $\mu$ g/L at 2 consecutive visits, whichever comes first.
- <sup>3</sup> Hematology: Hemoglobin, total WBC count, ANC, MCV, and platelet count.
- Blood chemistry: Total protein, GGT, glucose, bilirubin (total, direct, and indirect), AST, ALT, albumin, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, zinc. and CRP.
- The results obtained at screening for blood chemistry, physical examination, and urinalysis are considered to be the baseline results. These tests are not repeated at Day 0.
- <sup>6</sup> A blood sample for DNA testing is to be taken only if DNA confirmation of a diagnosis of beta-thalassemia is not available at the time of screening.
- Urinalysis: pH, specific gravity, glucose, protein, ketones, blood, and (if indicated by the dipstick results), sediment microscopy. If there is blood in the urine or three or more "plus signs" for protein, samples must be sent for microscopy.
- <sup>8</sup> Hepatitis B, hepatitis C, and HIV.
- <sup>9</sup> Heart rate, blood pressure, and body temperature. At the time of these measurements, the child must be calm and not crying.
- For infants not yet able to stand upright, stature is measured as recumbent length.
- For TSAT and SF, the values obtained at the screening visit (not those obtained at baseline) are used for the eligibility criteria.
- Blood samples for the assessment of prolactin are taken pre-dose and at +1.5 h +/-5 minutes post-dose. The second set of samples are taken only from patients who are still in the study at Month 12; they are not taken from patients who are terminated before that time.
- Dosing: Deferiprone oral solution 80 mg/mL or matching placebo solution.

#### 4. Measurements and Evaluations

# 4.1 Efficacy Measurements

Efficacy is measured by monitoring levels of serum ferritin, transferrin saturation, and labile plasma iron.

# 4.1.1 Serum Ferritin (μg/L)

Ferritin is a protein that stores iron in a non-toxic form, transports it to areas where it is required, and releases it in a controlled manner, thereby acting as a buffer against iron deficiency and iron overload. It is mainly found in tissues, but small amounts are measured in the serum, where it can serve as an indirect but easily measurable marker of the total amount of iron stored in the body. (Drawbacks of using it as a marker include lack of specificity, as disorders other than iron overload can cause large amounts of ferritin to be released into the circulation, and inter-patient variability.) Levels of serum ferritin above 1000 ng/mL are often considered to be associated with iron toxicity. In young children who have only recently begun an RBC transfusion regimen, it takes some time for this level to be reached, but in the absence of chelation it inevitably is reached.

Serum ferritin is measured at each visit, and the time to reach a level  $\geq 1000~\mu g/L$  will be compared between the treatment arms. Patient is to be withdrawn from the study when they attain a serum ferritin level  $\geq 1000~\mu g/L$  at 2 consecutive visits provided that the child has had no signs of infection in the previous 7 days and that CRP level is not greater than 20% higher than the normal range for the patient's age.

# 4.1.2 Transferrin Saturation (%)

Transferrin is a protein that combines with iron and transports it to where iron is required. When its capacity to bind incoming iron is exceeded, excess iron circulates as free non-transferrin-bound iron (NTBI) and is taken up by tissues where it can cause cell and organ damage. Transferrin saturation, defined as the percentage of the iron-binding sites of transferrin that are already occupied, is easily measured and hence serves as a marker for NTBI. High levels of transferrin saturation are associated with iron toxicity. As this measure is highly variable, the blood samples for its assessment are to be collected at approximately the same time of day and at approximately the same amount of time after the last dose of study medication, in an attempt to decrease variability as much as possible.

Transferrin saturation is measured at each visit, and the time to reach a level  $\geq$  60% will be compared between the treatment arms.

# 4.1.3 Labile Plasma Iron (μM)

Labile plasma iron is a component of NTBI, and is considered the most toxic form of iron since it acts as a catalyst in the formation of harmful free hydroxyl radicals which can damage cellular DNA,

proteins, and membrane lipids. High levels of this form of iron may be found in individuals with conditions of iron overload. As this measure is highly variable, the blood samples for its assessment are to be collected at approximately the same time of day and at approximately the same amount of time after the last dose of study medication, in an attempt to decrease variability as much as possible.

Labile plasma iron is measured at each visit, and the time to reach a level  $\geq 0.6 \mu M$  will be compared between the treatment arms.

# 4.2 Safety Measurements

# 4.2.1 Medical Events, Adverse Events, and Serious Adverse Events

Refer to section 7.2.1 of the LA55-0417 study protocol for the definitions of medical events, adverse events, and serious adverse events.

# 4.2.2 Laboratory Measurements

Analyses are performed at a central laboratory, with the exception of the weekly or biweekly hematology assessments which may be performed at a local laboratory. Investigators interpret each report promptly (preferably within 24 hours) and document their review by signing or initialing and dating it. Any laboratory values that fall outside a clinically accepted range, or that differ significantly from previous values, are assessed for clinical significance, and are marked by the investigator as either "CS" (clinically significant) or "NCS" (not clinically significant). Any clinically significant abnormalities or changes that are not part of a larger medical condition that is already recorded are further explained on the laboratory report and documented as an adverse event in the eCRF.

Samples for laboratory safety assessments are taken at the time points indicated below. If a patient withdraws from the study, the End of Study procedures are to be performed at an early termination visit.

| Hematology: Hemoglobin, total WBC count, ANC, MCV, and platelet count | Screening and weekly after start of dosing up to Month 6 visit, then biweekly until Month 12 or early termination from the study |
|---|---|
| Blood chemistry: Total protein, GGT, fasting glucose, bilirubin (total, direct, and indirect), AST, ALT, albumin, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, zinc, and C-reactive protein (CRP) | Screening and Months 1, 3, 6, 9, and 12 (or end of study) |

| <b>Urinalysis:</b> pH, specific gravity, glucose, protein, ketones, blood, and (if indicated by the dipstick results), sediment microscopy. If there is blood in the urine or three or more "plus signs" for protein, samples must be sent for microscopy. | Screening and Month 12 (or end of study) |
|---|---|
| Serology: Hepatitis B, hepatitis C, HIV | Screening |
| Other: Prolactin | Baseline and Month 12 |

# 4.2.3 Physical Examinations

Physical examination consists of an examination of head, ears, eyes, nose, throat and neck, respiratory system, cardiovascular system, gastrointestinal system, musculoskeletal system, neurological systems (central and peripheral), and skin, nails, hair, and scalp. It is to be performed at screening and at Months 1, 3, 6, 9, and 12 (or end of study). Any clinically significant abnormalities noted prior to the screening visit are recorded as medical history, any noted between screening and the first dose of study medication is recorded as medical events, and any that are noted post–Dose 1 are recorded as AEs.

The growth parameters of body weight and height (or length, in infants not yet able to stand upright) which are separate safety endpoints, are measured at each post-screening visit.

# 4.2.4 Vital Signs

Resting heart rate, resting blood pressure, and body temperature are taken. ("Resting" implies that the child must be calm and not crying.) Blood pressure should always be measured after a minimum 3-minute resting period, and using the same arm each time if possible. Systolic and diastolic blood pressures are to be recorded from one measurement.

Vital signs are measured at each site visit. Clinically significant out-of-range values for vital signs are reported as AEs.

### 4.2.5 Concomitant Medications

The following information about prior and concomitant medications are recorded:

- All medications used within the 3 months prior to baseline
- Any medications that the patient continues to take during the study
- Any medications that the patient starts to take during the study

The name, dose, route, frequency, indication, and stop and start dates of all medications used during the study must be noted in the source documents and CRFs, as well as whether or not the medication was used to treat an AE.

Information on concurrent medications are obtained at every site visit.

### 5. Statistical Analysis

A two-sided p-value of 0.05 will be used as the significance level for the determination of statistical significance in all statistical tests.

All statistical analyses of efficacy and safety data will be performed using SAS (version 9.4 or higher) on the Windows operating system.

## 5.1 Study Populations

# 5.1.1 Intent-to-Treat Population

The intent-to-treat (ITT) population will be composed of patients who were randomized, have received at least one dose of study medication, and have had at least one post-baseline measurement on the efficacy variables. All efficacy endpoints will be analyzed for the ITT population, which represents the primary analysis population.

# **5.1.2** Per Protocol Population

The per protocol (PP) population will represent the secondary analysis population, and will be composed of the same patients as in the intent-to-treat (ITT) population without major protocol deviations. Patients with major protocol deviation(s) will be determined before the database is locked. The efficacy endpoints will be analyzed for this population as well.

# **5.1.3** Safety Population

The safety population will be composed of patients who have received at least one dose of study medication.

### 5.2 Efficacy Endpoints

# 5.2.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the percentage of patients who still have a serum ferritin level  $< 1000 \,\mu\text{g/L}$  at Month 12.

# **5.2.2** Secondary Efficacy Endpoints

The secondary efficacy endpoints are:

- The percentage of patients whose serum ferritin level is still less than 1000 μg/L at each visit
- The percentage of patients whose LPI value is still less than 0.6 µM at each visit
- The percentage of patients whose TSAT value is still less than 60% at each visit
- Time to reach a serum ferritin level  $\geq 1000 \,\mu\text{g/L}$  (Note: a patient is to be withdrawn from the study only if the repeated serum ferritin level is  $\geq 1000 \,\mu\text{g/L}$ .)
- Time to reach an LPI value  $\geq 0.6 \mu M$
- Time to reach a TSAT value  $\geq 60\%$

### 5.3 Safety Endpoints

The safety endpoints are:

- Adverse events (AEs): Frequency, intensity, time to onset, duration, and relatedness to study drug
- Serious adverse events (SAEs): Frequency, intensity, time to onset, duration, and relatedness to study drug
- Number of discontinuations due to AEs
- Growth parameters: Weight, height, and height velocity, as classified using the Z-score system
- Change in prolactin level from baseline to Month 12

# 5.4 Patient Disposition and Drug Exposure

The numbers of patients who were screened, randomized, exposed to the study medication, who completed the study, and who withdrew from the study (along with reasons for withdrawals) will be presented.

### 5.5 Patient Characteristics

Patient characteristics at baseline, including demographics, will be summarized with descriptive statistics for continuous variables and with frequency tables for categorical variables. Medical history will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.0 or higher.

### 5.6 Analysis of Efficacy

The percentage of patients who have not reached levels of LPI  $\geq$  0.6  $\mu$ M, TSAT  $\geq$  60%, or SF  $\geq$  1000  $\mu$ g/L will be compared between the two treatment groups at each monthly time point as well as at the end of study, using the Fisher's exact test. (Note: the repeated SF value will be used to determine this for those patients whose SF is  $\geq$  1000  $\mu$ g/L.)

The effect of baseline value on each of the 3 efficacy endpoints will be examined in a covariate analysis. As an example for serum ferritin, the following SAS code of MIXED procedure will be used to produce the differences in Least Squares (LS) Mean of change in serum ferritin at Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 between deferiprone and placebo groups and the corresponding 95% confidence intervals.

```
proc mixed data=sf;
 class patient base sf treat month;
 model sf change = base sf treat month treat*month /
 noint solution ddfm=kr;
  repeated month / Patient=patient(treat) type=ar(1);
  lsmeans treat*month;
 estimate 'Deferiprone - Placebo at Month 1'
            treat 1 -1
            treat*month 1 0 0 0 0 0 0 0 0 0 0
                        -1 0 0 0 0 0 0 0 0 0 0 0 0 / cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 2'
            treat 1 -1
            treat*month 0
                            1 0 0 0 0 0 0 0 0 0
                         0 -1 0 0 0 0 0 0 0 0 0 0 / cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 3'
            treat 1 -1
           treat*month 0 0 1 0 0 0 0 0 0 0 0
                         0 0 -1 0 0 0 0 0 0 0 0 0 0 cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 4'
            treat 1 -1
                         0 0 0 1 0 0 0 0 0 0 0
            treat*month
                         0 0 0 -1 0 0 0 0 0 0 0 0 0 cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 5'
            treat 1 -1
            treat*month 0 0 0 0 1 0 0 0 0 0 0
                         0 0 0 0 -1 0 0 0 0 0 0 0 / cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 6'
            treat 1 -1
            treat*month
                         0 0 0 0 0 1 0 0 0 0 0
                         0 0 0 0 0 -1 0 0 0 0 0 0 0 cl alpha=0.05;
```

```
estimate 'Deferiprone - Placebo at Month 7'
           treat 1 -1
           treat*month 0 0 0 0 0 0 1 0 0 0 0
                        0 0 0 0 0 0 -1 0 0 0 0 0 / cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 8'
           treat 1 -1
                        0 0 0 0 0 0 0 1 0 0 0
           treat*month
                        0 0 0 0 0 0 0 -1 0 0 0 0/ cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 9'
           treat 1 -1
           treat*month 0 0 0 0 0 0 0 1 0 0 0
                        0 0 0 0 0 0 0 0 -1 0 0 0/ cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 10'
           treat 1 -1
           treat*month 0 0 0 0 0 0 0 0 1 0 0
                        0 0 0 0 0 0 0 0 0 -1 0 0/ cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 11'
           treat 1 -1
           treat*month 0 0 0 0 0 0 0 0 0 1 0
                        0 0 0 0 0 0 0 0 0 0 -1 0/ cl alpha=0.05;
 estimate 'Deferiprone - Placebo at Month 12'
           treat 1 -1
           treat*month 0 0 0 0 0 0 0 0 0 0 1
                        0 0 0 0 0 0 0 0 0 0 0 -1/ cl alpha=0.05;
run;
```

A Kaplan-Meier survival curve for the time to reach a serum ferritin level  $\geq$  1000 µg/L, an LPI value  $\geq$  0.6 µM, or a TSAT value  $\geq$  60% will be generated for the two treatment groups. Log-rank test will be used for comparing the two survival curves for each of the 3 efficacy endpoints.

As an example, for serum ferritin, the following SAS code of LIFETEST procedure will be used to compare the two survival curves. A variable status is the censoring indicator. A status of 1 indicates an event time when a serum ferritin level reaches  $\geq 1000~\mu g/L$  and a status of 0 indicates the event of serum ferritin level  $\geq 1000~\mu g/L$  has not occurred by the end of the study.

```
proc lifetest data=sf method=km plot=(s) graphics;
  time month*status(0);
  strata treat;
run;
```

Trend analysis over time for LPI, TSAT, and SF measures will be performed to compare the rate of change per month in these measures between the two treatment groups. As an example, for serum ferritin, the following SAS code of MIXED procedure will be used to compare the two slopes between the two treatment groups:

```
proc mixed data=sf;
  class treat patient;
  model sf = treat month treat*month / noint solution;
  repeated / type=ar(1) Patient=patient(treat);
  estimate 'Slope for deferiprone' month 1 treat*month 1 0;
  estimate 'Slope for placebo' month 1 treat*month 0 1;
  estimate 'Slope for deferiprone minus placebo' treat*month 1 -1;
  run;
```

## 5.7 Analysis of Safety

Descriptive statistics (mean, standard deviation, minimum, and maximum) will be produced for continuous variables, and frequency tables will be produced for discrete variables by treatment group. Summaries of adverse events and serious adverse events will be produced by treatment group. Shift tables will be generated for comparing the screening/baseline values and end of study values of the relevant measures.

The following safety data will be summarized by treatment group:

- Adverse events (AEs), adverse drug reactions (ADRs), serious adverse events (SAEs), and serious adverse drug reactions (SADRs)
- Number of discontinuations due to AEs
- Hematology assessments
- Biochemistry assessments
- Urinalysis
- Vital signs
- Prior and concomitant medications

Prolactin is measured at baseline and Month 12. The change in prolactin level from baseline to Month 12 will be compared between the two treatment groups using an ANCOVA model with baseline value as a covariate and treatment as the main factor.

#### 5.7.1 AEs and SAEs

Adverse events (AEs) are coded using MedDRA version 23.0 or higher. In counting the number of patients who experienced each AE, any patients who experienced the same AE multiple times will be counted only once for the corresponding preferred term (PT). Similarly, any patients who experienced multiple AEs within the same system organ class (SOC) will be counted only once for that SOC. AEs will be tabulated alphabetically by SOC; and within each SOC, the PTs will be presented alphabetically. In tables that present the incidence of AEs by severity, seriousness, and relation to study

medication, any patients with multiple events coded to a given PT or SOC will be counted only once for that PT or SOC according to the most severe event, the most serious event, or the event with the closest relationship to study medication.

AEs will be summarized for the total number of AEs, the total number and percent of patients who experienced at least one AE, and the total number and percent of patients who experienced an AE within each SOC (and each PT within an SOC). A p-value comparing the percentages of each AE among treatment groups will be calculated by using Fisher's exact test.

The incidences of AEs, SAEs, adverse drug reactions (ADRs), and serious ADRs (SADRs) will be tabulated by treatment group. The relationship to study medication for AEs will be tabulated by treatment group.

A listing of SAEs and a listing of withdrawals due to AEs with time to withdrawal will be produced. Any deaths will be listed separately and discussed in narratives.

### 5.7.2 Number of discontinuations due to AEs

The percent of patients who have been withdrawn for the study due to AEs will be compared between the two treatment groups using Fisher's exact test.

# 5.7.3 Hematology and biochemistry

Hematology and biochemistry data will be summarized by using descriptive statistics at each assessment by treatment group. Change from baseline to each follow-up assessment will also be summarized by using descriptive statistics by treatment group. The data listings of patients who have abnormal values as well as patients who have clinically significant values will be produced for each parameter. The number (%) of patients who have ALT  $> 2 \times ULN$ , 3 x ULN, and 5 x ULN during the study will be compared between the two treatment groups.

### 5.7.4 Urinalysis

Urinalysis assessments consist of pH, specific gravity, glucose, protein, ketones, blood, and (if indicated by the dipstick results), sediment microscopy. If there is blood in the urine or three or more "plus signs" for protein, samples must be sent for microscopy. Clinically significant laboratory values for urinalysis are reported as AEs.

## 5.7.5 Vital signs

Temperature, resting heart rate, and diastolic and systolic blood pressures will be summarized using descriptive statistics at each assessment by treatment group. Change from baseline to each follow-up assessment will be also summarized using descriptive statistics by treatment group.

#### 5.7.6 Prior and concomitant medications

Prior and concomitant medications are summarized using the WHO Drug Dictionary (WHO-DD) version B2 (March 2018).

#### 5.7.7 Time to withdrawal

A Kaplan-Meier survival curve for the time to be withdrawn from the study will be generated for the two treatment groups. The Log-rank test will be used for comparing the two survival curves.

# 5.7.8 Height and weight

For height (cm) and weight (kg), the change from baseline to last assessment will be compared between the two treatment groups using an ANCOVA model with baseline value as a covariate and treatment as the main factor. The rate of change in height will be assessed using regression analysis.

Child growth standards for 2007 are available at the WHO website <a href="https://www.who.int/childgrowth/standards/en/">https://www.who.int/childgrowth/standards/en/</a>. This site provides mean and standard deviation for height from 0 to 5 years old by day for males and females. It has mean and standard deviation for height from 5 to 19 years old by month for male and female and for weight from 5 to 10 years old by month for males and females.

Z scores will be calculated by matching sex and age in days until 5 years old and by matching sex and age in months from 5 to 10 years old as follows:

(Observed data from LA55 – Mean from WHO data) / (Standard deviation from WHO data)

The change from baseline to last assessment in Z score will be compared between the two treatment groups using an ANCOVA model with baseline value as a covariate and treatment as the main factor.

### Impact of COVID-19 on the primary efficacy endpoints

Sensitivity analyses may be performed, if warranted, by excluding data that might have been impacted by COVID-19.

#### **SUMMARY TABLES AND FIGURES**

Summary tables and figures are numbered following ICH structure.

Note: The final numberings for tables and/or figures in the clinical study report can be changed if more tables and/or figures are made in the addition to those in the SAP.

#### **TABLES**

### 14.1 Patient disposition, demographics, and baseline data

- Table 14.1.1 Patient disposition
- Table 14.1.2 Number of patients by study site
- Table 14.1.3 Number of patients in safety, ITT, and PP populations
- Table 14.1.4 Reasons for not completing the study
- Table 14.1.5 Demographics data
- Table 14.1.6 Medical history
- Table 14.1.7 Serum ferritin, LPI, and TSAT at baseline

### 14.2 Efficacy analyses

# 14.2.1 Serum ferritin (μg/L)

- Table 14.2.1.1 Serum ferritin (µg/L) at each assessment ITT population
- Table 14.2.1.1a Serum ferritin (µg/L) at each assessment PP population
- Table 14.2.1.2 Change in serum ferritin (μg/L) from baseline at each follow-up assessment ITT population
- Table 14.2.1.2a Change in serum ferritin ( $\mu$ g/L) from baseline at each follow-up assessment PP population
- Table 14.2.1.3 LS Means for change in serum ferritin ( $\mu g/L$ ) from ANCOVA model at each follow-up assessment ITT population
- Table 14.2.1.3a LS Means for change in serum ferritin ( $\mu g/L$ ) from ANCOVA model at each follow-up assessment ITT population
- Table 14.2.1.4 Trend analysis for serum ferritin (µg/L) over time ITT population
- Table 14.2.1.4a Trend analysis for serum ferritin ( $\mu$ g/L) over time PP population
- Table 14.2.1.5 Percent of patients who had serum ferritin < 1000 μg/L at each assessment ITT population
- Table 14.2.1.5a Percent of patients who had serum ferritin < 1000 μg/L at each assessment PP population

### 14.2.2 Labile plasma iron (μM)

Table 14.2.2.1 LPI (μM) at each assessment – ITT population

- Table 14.2.2.1a LPI ( $\mu$ M) at each assessment PP population
- Table 14.2.2.2 Change in LPI (µM) from baseline at each follow-up assessment ITT population
- Table 14.2.2.2a Change in LPI (μM) from baseline at each follow-up assessment PP population
- Table 14.2.2.3 LS Means for change in LPI ( $\mu$ M) from ANCOVA model at each follow-up assessment ITT population
- Table 14.2.2.3a LS Means for change in LPI ( $\mu$ M) from ANCOVA model at each follow-up assessment PP population
- Table 14.2.2.4 Trend analysis for LPI (μM) over time ITT population
- Table 14.2.2.4a Trend analysis for LPI (μM) over time PP population
- Table 14.2.2.5 Percent of patients who had LPI < 0.6 μM at each assessment ITT population
- Table 14.2.2.5a Percent of patients who had LPI  $\leq 0.6 \,\mu\text{M}$  at each assessment PP population

#### 14.2.3 Transferrin saturation (%)

- Table 14.2.3.1 TSAT (%) at each assessment ITT population
- Table 14.2.3.1a TSAT (%) at each assessment PP population
- Table 14.2.3.2 Change in TSAT (%) from baseline at each follow-up assessment ITT population
- Table 14.2.3.2a Change in TSAT (%) from baseline at each follow-up assessment PP population
- Table 14.2.3.3 LS Means for change in TSAT (%) from ANCOVA model at each follow-up assessment ITT population
- Table 14.2.3.3a LS Means for change in TSAT (%) from ANCOVA model at each follow-up assessment PP population
- Table 14.2.3.4 Trend analysis for TSAT (%) over time ITT population
- Table 14.2.3.4a Trend analysis for TSAT (%) over time PP population
- Table 14.2.3.5 Percent of patients who had TSAT < 60% at each assessment ITT population
- Table 14.2.3.5a Percent of patients who had TSAT < 60% at each assessment PP population

#### 14.3 Safety analyses

#### 14.3.1 Adverse events

- Table 14.3.1.1 Overall summary of adverse events
- Table 14.3.1.2 Adverse events

- Table 14.3.1.3 Most common Adverse Events >= 5 percent
- Table 14.3.1.4 Adverse events with the maximum severity/intensity
- Table 14.3.1.5 Adverse drug reactions
- Table 14.3.1.6 Most common Adverse drug reactions >= 5 percent
- Table 14.3.1.7 Adverse drug reaction with the maximum severity/intensity
- Table 14.3.1.8 Serious adverse events
- Table 14.3.1.9 Serious adverse events with the maximum severity/intensity
- Table 14.3.1.10 Serious adverse drug reactions
- Table 14.3.1.11 Serious adverse drug reactions with the maximum severity/intensity
- Table 14.3.1.12 Adverse events by relatedness to study medication
- Table 14.3.1.13 Adverse events event count and rate

### 14.3.2 Vital signs

- Table 14.3.2.1 Temperature (C) Heart rate at each assessment
- Table 14.3.2.2 Change in temperature (C) from baseline at each follow-up assessment
- Table 14.3.2.3 Heart rate (bpm) at each assessment
- Table 14.3.2.4 Change in heart rate (bpm) from baseline to each follow-up assessment
- Table 14.3.2.5 Diastolic blood pressure (mmHg) at each assessment
- Table 14.3.2.6 Change in diastolic blood pressure (mmHg) from baseline at each follow-up assessment
- Table 14.3.2.7 Systolic blood pressure (mmHg) at each assessment
- Table 14.3.2.8 Change in systolic blood pressure (mmHg) from baseline at each follow-up assessment

#### 14.3.3 Height

- Table 14.3.3.1 Height (cm) at each assessment
- Table 14.3.3.2 Change in height (cm) from baseline to at each follow-up assessment
- Table 14.3.3.3 LS Means for change in height (cm) from ANCOVA model at Month 12
- Table 14.3.3.4 Trend analysis for height (cm) over time
- Table 14.3.3.5 Z score analysis for height (cm)

### 14.3.4 Weight

- Table 14.3.4.1 Weight (kg) at each assessment
- Table 14.3.4.2 Change in weight (kg) from baseline to at each follow-up assessment
- Table 14.3.4.3 LS Means for change in weight (kg) from ANCOVA model at Month 12

Table 14.3.4.4 Trend analysis for weight (kg) over time

Table 14.3.4.5 Z score analysis for weight (kg)

#### 14.3.5 Concomitant medications

Table 14.3.4.1 Concomitant medications

### 14.3.6 Laboratory data

#### 14.3.6.1 Hematology

Table 14.3.6.1.1 Hematology data at each assessment

Table 14.3.6.1.2 Change in hematology data from baseline to each follow-up assessment

Table 14.3.6.1.3 Shift table for hematology data: deferiprone group

Table 14.3.6.1.4 Shift table for hematology data: placebo group

### 14.3.6.2 Biochemistry

Table 14.3.6.2.1 Biochemistry data at each assessment

Table 14.3.6.2.2 Change in biochemistry data from baseline to at each follow-up assessment

Table 14.3.6.2.3 Shift table for biochemistry data: deferiprone group

Table 14.3.6.2.4 Shift table for biochemistry data: placebo group

Table 14.2.6.2.5 Percent of patients who had ALT > 2 x ULN, 3 x ULN, or 5 x ULN during the study

Table 14.2.6.2.6 Percent of patients who had AST > 2 x ULN, 3 x ULN, or 5 x ULN during the study

#### 14.3.7 Prolactin

Table 14.3.7.1 Prolactin at each assessment

Table 14.3.7.2 Change in prolactin from pre-dose to Month 12

Table 14.3.7.3 LS Means of change in prolactin from pre-dose to Month 12 from the ANCOVA model

### 14.4 Other analyses

Table 14.4.1 Compliance (%) at each assessment

Table 14.4.2 Overall mean of transfusional iron input (mg/kg/day) during the study

Table 14.4.3 Overall mean of total daily dose (mg/kg/day) during the study

Table 14.1.4 Patient exposure to study medication

Table 14.1.5 Duration of study drug exposure

### **FIGURES**

## 14.2 Efficacy

- Figure 14.2.1 Mean line graph for serum ferritin over time
- Figure 14.2.2 Mean line graph for LPI over time
- Figure 14.2.3 Mean line graph for TSAT over time
- Figure 14.2.4 Mean line graph for change from baseline in serum ferritin over time
- Figure 14.2.5 Mean line graph for change from baseline in LPI over time
- Figure 14.2.6 Mean line graph for change from baseline in TSAT over time
- Figure 14.2.7 Kaplan-Meier survival curve for the time to reach serum ferritin level ≥ 1000 μg/L
- Figure 14.2.8 Kaplan-Meier survival curve for the time to reach LPI value ≥ 0.6 μM
- Figure 14.2.9 Kaplan-Meier survival curve for the time to reach TSAT value ≥ 60%

#### 14.3 Safety

### 14.3.1 Hematology

- Figure 14.3.1.1 Mean line graph for the hematology data over visit
- Figure 14.3.1.2 Proportion of patients with abnormal hematology data at each assessment
- Figure 14.3.1.3 ANC graphs for patients with neutropenia
- Figure 14.3.1.4 ANC graphs for patients with agranulocytosis

### 14.3.2 Biochemistry

- Figure 14.3.2.1 Mean line graph for the biochemistry data over visit
- Figure 14.3.2.2 Proportion of patients with abnormal biochemistry data at each assessment

#### 16.1.9 Documents of Statistical Methods

- SAS output 16.1.9.1 Kaplan-Meier survival analysis for the time to reach serum ferritin level ≥ 1000 µg/L
- SAS output 16.1.9.2 Kaplan-Meier survival analysis for the time to reach LPI value  $\geq 0.6 \mu M$
- SAS output 16.1.9.3 Kaplan-Meier survival analysis for the time to reach TSAT value  $\geq 60\%$
- SAS output 16.1.9.4 Kaplan-Meier survival analysis for the time to be withdrawn from the study

#### **DATA LISTINGS**

Data listings are numbered following ICH structure.

Note: The final numberings for Patient data listings in the clinical study report can be changed if more Patient data listings are made in the addition to those in the SAP.

### 16.2.1 Discontinued patients

- 16.2.1.1 Listing of disposition
- 16.2.1.2 Listing of withdrawals due to AEs

# 16.2.2 Protocol deviation

- 16.2.2.1 Listing of assessed protocol deviations
- 16.2.2.2 Listing of protocol deviations monitoring plan (Appendix C)

# 16.2.3 Patients excluded from efficacy

16.2.3.1 Listing of assignment of patients to analysis sets

## 16.2.4 Demographic data

16.2.4.1 Listing of demographics

## 16.2.5 Compliance\_Drug concentration data

16.2.5.1 Listing of compliance

### 16.2.6 Individual efficacy response data

- 16.2.6.1 Listing of labile plasma iron (LPI)
- 16.2.6.2 Listing of serum ferritin (SF)
- 16.2.6.3 Listing of transferrin saturation (TSAT)

### 16.2.7 Adverse events

- 16.2.7.1 Listing of medical events
- 16.2.7.2 Listing of adverse events
- 16.2.7.3 Listing of serious adverse events

#### 16.2.8 Individual lab measurements by patient

- 16.2.8.1 Listing of hematology
- 16.2.8.1a Listing of patients who have had abnormal values in hematology
- 16.2.8.1b Listing of patients who have had clinically significant values in hematology
- 16.2.8.2 Listing of urinalysis
- 16.2.8.3 Listing of serology
- 16.2.8.4 Listing of biochemistry
- 16.2.8.4a Listing of patients who have had abnormal values in biochemistry

16.2.8.4b Listing of patients who have had clinically significant values in biochemistry 16.2.8.5 Listing of prolactin

# **16.2.9 Other measurements**

- 16.2.9.1 Listing of informed consent / Assent form
- 16.2.9.2 Listing of primary diagnosis
- 16.2.9.3 Listing of medical history
- 16.2.9.4 Listing of randomization
- 16.2.9.5 Listing of vital signs
- 16.2.9.6 Listing of physical examination
- 16.2.9.7 Listing of transfusion
- 16.2.9.8 Listing of exposure
- 16.2.9.9 Listing of concomitant medications

### **TABLE SHELLS**

The following table shells provide a framework for the display of data from this study. These tables may not be designed exactly as shown in the shells, but are intended to reflect the general layout of the data that will be included in the clinical study report.

Note that 'c' in the table shells indicates an alphanumeric character and 'x' indicates a number from 0 to 9.

# 14.1 Patient disposition, demographics, and baseline data

Table 14.1.1 Patient disposition

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|------------|-------------|-----------|----------------------------------|
| Randomized | xxx | xxx | |
| Exposed | xxx (xx%) | xxx (xx%) | 0.xxxx |
| Completed | xxx (xx%) | xxx (xx%) | 0.xxxx |
| Withdrawn | xxx (xx%) | xxx (xx%) | 0.xxxx |

Data source: 16.2.1.1 Listing of disposition

Table 14.1.2 Number of patients by study site

| Country | Site | Deferiprone | Placebo | Total |
|-----------|-------|-------------|---------|-------|
| Egypt | 003 | XX | XX | xx |
| | 004 | XX | XX | XX |
| | 005 | XX | XX | xx |
| Indonesia | 006 | XX | XX | xx |
| | Total | XX | XX | XX |

Data source: 16.2.4.1 Listing of demographics

Table 14.1.3 Number of patients in safety, ITT, and PP populations

| | | Deferiprone | Placebo |
|-------------------|----------------|-------------|---------|
| Safety population | | xx | XX |
| | Serum ferritin | XX | XX |
| ITT population | LPI | XX | XX |
| | TSAT | XX | XX |
| | Serum ferritin | XX | XX |
| PP population | LPI | XX | XX |
| | TSAT | XX | XX |

Data source: 16.2.3.1 Listing of assignment of patients to analysis sets

Table 14.1.4 Reasons for not completing the study

| | | Deferiprone | Placebo | Total |
|-------------------------------|--------|-------------|----------|----------|
| | | n (%) | n (%) | n (%) |
| N | | xx (100) | xx (100) | xx (100) |
| Reason: | Detail | | | |
| Adverse event | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Withdrawal by parent/guardian | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Lost to follow-up | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Physician decision | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Protocol deviation | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Lack of efficacy | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Other | Cccc | xx (xx) | xx (xx) | xx (xx) |
| | Cccc | xx (xx) | xx (xx) | xx (xx) |
| Total | | xx (xx) | xx (xx) | xx (xx) |

Data source: 16.2.1.1 Listing of disposition

Table 14.1.5 Demographics data

| | Deferiprone | Placebo | Total | |
|---|---|---|---|---|
| N | XX | xx | xx | p-value§ |
| Age (years): | | | | 0.xxxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | xx.x | xx.x | |
| Sex: n (%) | | | | 0.xxxx |
| Female | xx (xx) | xx (xx) | xx (xx) | |
| Male | xx (xx) | xx (xx) | xx (xx) | |
| Ethnic Origin: n (%) | | | | 0.xxxx |
| Hispanic/Latino | xx (xx) | xx (xx) | xx (xx) | |
| Not Hispanic/Latino | xx (xx) | xx (xx) | xx (xx) | |
| Racial Origin: n (%) | | | | 0.xxxx |
| Asian | xx (xx) | xx (xx) | xx (xx) | |
| American Indian or Alaska Native | xx (xx) | xx (xx) | xx (xx) | |
| Black or African American | xx (xx) | xx (xx) | xx (xx) | |
| Native Hawaiian or Other Pacific Islander | xx (xx) | xx (xx) | xx (xx) | |
| White | xx (xx) | xx (xx) | xx (xx) | |
| Other | xx(xx) | xx(xx) | xx(xx) | |

§T-test for age; Fisher's exact test for sex, ethnic origin, and racial origin Data source: 16.2.4.1 Listing of demographics
Table 14.1.6 Medical history

| | Deferiprone | | Placebo | | Total | |
|---|---|---|---|---|---|---|
| N | xx | | xx | | XX | |
| Illness/Event by | Resolved | ongoing | resolved | ongoing | resolved | ongoing |
| MedDRA Primary | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class and<br>Preferred Term | | | | | | |
| Cccccc | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Ceeece | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Ceeece | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Ceeece | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

Data source: 16.2.9.3 Listing of medical history

Table 14.1.7 Serum ferritin, LPI, and TSAT at baseline

| | Deferiprone | Placebo | |
|----------------|-----------------|-----------------|------------------|
| N | XX | XX | |
| | $Mean \pm SD$ | $Mean \pm SD$ | P-value (t-test) |
| | (Min, Max) | (Min, Max) | , , |
| Serum Ferritin | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | 0.xxxx |
| (µg/L) | (xxxx, xxxx) | (xxxx, xxxx) | |
| / | $x.xx \pm x.xx$ | $x.xx \pm x.xx$ | 0.xxxx |
| LPI (μM) | (x.xx, x.xx) | (x.xx, x.xx) | |
| | $xx \pm xx$ | $xx \pm xx$ | 0.xxxx |
| TSAT (%) | (xx, xx) | (xx, xx) | |

Data source: 16.2.6.2 Listing of serum ferritin (SF)

16.2.6.1 Listing of labile plasma iron (LPI)

16.2.6.3 Listing of transferrin saturation (TSAT)

Table 14.1.8 Serology data at baseline

| Positive result | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|---|---|---|---|
| Hepatitis B | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Hepatitis C | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| HIV | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

Data source: 16.2.8.3 Listing of serology

## 14.2 Efficacy Analyses

## 14.2.1 Serum Ferritin (μg/L)

Table 14.2.1.1 Serum ferritin ( $\mu$ g/L) at each assessment – ITT population

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Baseline | XX | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx (xxxx,xxxx)$ | 0.xxxx |
| Month 1 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 2 | xx | xxxx ± xxxx (xxxx,xxxx) | XX | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 3 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 4 | XX | xxxx ± xxxx (xxxx,xxxx) | XX | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 5 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 6 | xx | xxxx ± xxxx (xxxx,xxxx) | XX | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 7 | XX | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 8 | XX | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 9 | xx | xxxx ± xxxx (xxxx,xxxx) | XX | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 10 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 11 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx (xxxx,xxxx)$ | 0.xxxx |
| Month 12 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |

Data source: 16.2.6.2 Listing of serum ferritin (SF)

Note: Similar Table 14.2.1.1a will be made for PP population

Table 14.2.1.2 Change in serum ferritin ( $\mu g/L$ ) from baseline to each follow-up assessment – ITT population

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Month 1 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 2 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 3 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 4 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 5 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |
| Month 6 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 7 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 8 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 9 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 10 | xx | xxxx ± xxxx (xxxx,xxxx) | XX | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 11 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx \\ (xxxx,xxxx)$ | 0.xxxx |
| Month 12 | xx | xxxx ± xxxx (xxxx,xxxx) | xx | $xxxx \pm xxxx$ $(xxxx,xxxx)$ | 0.xxxx |

Data source: 16.2.6.2 Listing of serum ferritin (SF)

Note: Similar Table 14.2.1.2a will be made for PP population

Table 14.2.1.3 LS Means for change in serum ferritin (µg/L) from ANCOVA model at each followup assessment – ITT population

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | XX | XX | |
| | LS Mean ± SE | LS Mean ± SE | LS Mean ± SE | |
| Month 1 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 2 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 3 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 4 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 5 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 6 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 7 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 8 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 9 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 10 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 11 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |
| Month 12 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |

Data source: 16.2.6.2 Listing of serum ferritin (SF)
Note: Similar Table 14.2.1.3a will be made for PP population

Table 14.2.1.4 Trend analysis for serum ferritin (µg/L) over time – ITT population

| Rate of change per month | Deferiprone | Placebo | Deferiprone<br>minus Placebo | P-value |
|---|---|---|---|---|
| Mean ± SE | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | 0.xxxx |

Data source: 16.2.6.2 Listing of serum ferritin (SF)

Note: Similar Table 14.2.1.4a will be made for PP population

Table 14.2.1.5 Percent of patients who had serum ferritin  $\leq$  1000  $\mu g/L$  at each assessment - ITT population

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|----------|---------------|---------------|----------------------------------|
| Baseline | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 1 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 2 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 3 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 4 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 5 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 6 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 7 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 8 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 9 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 10 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 11 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 12 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

Data source: 16.2.6.2 Listing of serum ferritin (SF)

Note: Similar Table 14.2.1.5a will be made for PP population

## 14.2.2 Labile Plasma Iron (μM)

Table 14.2.2.1 LPI ( $\mu M$ ) each assessment – ITT population

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Baseline | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 1 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 2 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 3 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 4 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 5 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 6 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 7 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 8 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 9 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 10 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 11 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 12 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |

Data source: 16.2.6.1 Listing of labile plasma iron (LPI)

Note: Similar Table 14.2.2.1a will be made for PP population

Table 14.2.2.2 Change in LPI ( $\mu M$ ) from baseline to each follow-up assessment – ITT population

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Month 1 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 2 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 3 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 4 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 5 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 6 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 7 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 8 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 9 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 10 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 11 | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | xx | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |
| Month 12 | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | XX | $x.xx \pm x.xx (x.xx, x.xx)$ | 0.xxxx |

Data source: 16.2.6.1 Listing of labile plasma iron (LPI)

Note: Similar Table 14.2.2.1a will be made for PP population

Table 14.2.2.3 LS Means for change in LPI (µM) from ANCOVA model at each follow-up assessment – ITT population

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | XX | XX | |
| | LS Mean ± SE | LS Mean ± SE | LS Mean ± SE | |
| Month 1 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 2 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 3 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 4 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 5 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 6 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 7 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 8 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 9 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 10 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 11 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |
| Month 12 | $x.xx \pm x.xx$ | $x.xx \pm x,xx$ | $x.xx \pm x.xx$ | (x.xx, x.xx) |

Data source: 16.2.6.1 Listing of labile plasma iron (LPI)
Note: Similar Table 14.2.2.3a will be made for PP population

Table 14.2.2.4 Trend analysis for LPI ( $\mu M$ ) over time – ITT population

| Rate of change per month | Deferiprone | Placebo | Deferiprone<br>minus Placebo | P-value |
|---|---|---|---|---|
| Mean ± SE | $x.xx \pm x.xx$ | $x.xx \pm x.xx$ | $x.xx \pm x.xx$ | 0.xxxx |

Data source: 16.2.6.1 Listing of labile plasma iron (LPI)
Note: Similar Table 14.2.2.4a will be made for PP population

Table 14.2.2.5 Percent of patients who had LPI  $< 0.6 \mu M$  at each assessment – ITT population

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|----------|---------------|---------------|----------------------------------|
| Baseline | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 1 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 2 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 3 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 4 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 5 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 6 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 7 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 8 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 9 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 10 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 11 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 12 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

Data source: 16.2.6.1 Listing of labile plasma iron (LPI)
Note: Similar Table 14.2.2.5a will be made for PP population

## 14.2.3 Transferrin Saturation (%)

Table 14.2.3.1 TSAT (%) each assessment – ITT population

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Baseline | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 1 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 2 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 3 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 4 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 5 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 6 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 7 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 8 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 9 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 10 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 11 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 12 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |

Data source: 16.2.6.3 Listing of transferrin saturation (TSAT) Note: Similar Table 14.2.3.1a will be made for PP population

Table 14.2.3.2 Change in TSAT (%) from baseline to each follow-up assessment – ITT population

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Month 1 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 2 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 3 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 4 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 5 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 6 | XX | $xx.x \pm xx.x (xx.x, xx.x)$ | XX | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 7 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 8 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 9 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 10 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 11 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |
| Month 12 | xx | $xx.x \pm xx.x (xx.x, xx.x)$ | xx | $xx.x \pm xx.x (xx.x, x.xx)$ | 0.xxxx |

Data source: 16.2.6.3 Listing of transferrin saturation (TSAT) Note: Similar Table 14.2.3.2a will be made for PP population

Table 14.2.3.3 LS Means for change in TSAT (%) from ANCOVA model at each follow-up assessment – ITT population

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | XX | XX | |
| | LS Mean ± SE | LS Mean ± SE | LS Mean ± SE | |
| Month 1 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 2 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 3 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 4 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 5 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 6 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 7 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 8 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 9 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 10 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 11 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |
| Month 12 | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | (xx.x, xx.x) |

Data source: 16.2.6.3 Listing of transferrin saturation (TSAT) Note: Similar Table 14.2.3.3a will be made for PP population

CONFIDENTIAL

Table 14.2.3.4 Trend analysis for TSAT (%) over time – ITT population

| Rate of change per month | Deferiprone | Placebo | Deferiprone<br>minus Placebo | P-value |
|---|---|---|---|---|
| Mean ± SE | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | 0.xxxx |

Data source: 16.2.6.3 Listing of transferrin saturation (TSAT) Note: Similar Table 14.2.3.4a will be made for PP population

Table 14.2.3.5 Percent of patients who had TSAT < 60% at each assessment – ITT population

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|----------|---------------|---------------|----------------------------------|
| Baseline | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 1 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 2 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 3 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 4 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 5 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 6 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 7 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 8 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 9 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 10 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 11 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| Month 12 | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

Data source: 16.2.6.3 Listing of transferrin saturation (TSAT) Note: Similar Table 14.2.3.5a will be made for PP population

## 14.3 Safety analyses

#### 14.3.1 Adverse events

Table 14.3.1.1 Overall summary of adverse events

| | Deferiprone | Placebo | |
|---|---|---|---|
| N | xxx | xxx | P-<br>value |
| Number of patients experiencing at least one AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one severe AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one serious AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patients experiencing at least one related* AE | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patient deaths | xx (xx%) | xx (xx%) | 0.xxxx |
| Number of patient withdrawals due to AEs | xx (xx%) | xx (xx%) | 0.xxxx |

<sup>\*</sup>Includes possibly, probably, and definitely related. Worst case scenario of causality between the investigator and company's assessment.

Data source: 16.2.7.2 Listing of adverse events

Table14.3.1.2 Adverse events

| | Deferiprone<br>(N=xx) | Placebo<br>(N=xx) | Fisher's |
|---|---|---|---|
| | Exposure (Patient-years):x.xx | | exact test |
| | Total Events: xxx | Total Events: xxx | |
| System Organ Class<br>Preferred Term | n Patients (%) | n Patients (%) | p-value |
| CCCCCC | x (x.x) | x (x.x) | 0.xxxx |
| Cecee | x (x.x) | x (x.x) | 0.xxxx |
| Ccccc | x (x.x) | x (x.x) | 0.xxxx |
| Cecee | x (x.x) | x (x.x) | 0.xxxx |

Data source: 16.2.7.2 Listing of adverse events

Note: Similar Table 14.3.1.2 to Table 14.3.1.11 will be produced.

Table 14.3.1.12 Adverse events by causality

| | | Deferiprone<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| System Organ Class<br>Preferred Term | Relatedness<br>(worst case) | Patients reporting (n=xx) | Patients reporting (n=xx) |
| CCCCCCC | | x (x.x) | x (x.x) |
| ccccc | Not Related | x (x.x) | x (x.x) |
| | Related* | x (x.x) | x (x.x) |
| ccccc | Not Related | x (x.x) | x (x.x) |
| | Related* | x (x.x) | x (x.x) |

<sup>\*</sup>Possibly, Probably, or Definitely Related Data source: 16.2.7.2 Listing of adverse events

Table 14.3.1.13 Adverse events – event count and rate

| | Deferiprone (N=xx) | Placebo<br>(N=xx) |
|---|---|---|
| | Exposure (Patient-years):x.xx | Exposure (Patient-years):x.xx |
| | Total Events (Rate/100 patient- years): xx (x.xx) | Total Events (Rate/100 patient- years): xx (x.xx) |
| System Organ Class Preferred Term | xx (x.xx) | (x.xx) |
| CCCCCC | xx (x.xx) | xx (x.xx) |
| Ccccc | xx (x.xx) | xx (x.xx) |
| Ccccc | xx (x.xx) | xx (x.xx) |
| Cecece | xx (x.xx) | xx (x.xx) |

Data source: 16.2.7.2 Listing of adverse events

## 14.3.2 Vital signs

Table 14.3.2.1 Temperature (C) at each assessment

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Baseline | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 1 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 2 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 3 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 4 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 5 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 6 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 7 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 8 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 9 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 10 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 11 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 12 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.9.5 Listing of vital signs

Note: Similar Tables 14.3.2.3, 14.3.2.5, and 14.3.2.7 for heart rate, diastolic blood pressure, and

systolic blood pressure will be produced, respectively.

Table 14.3.2.2 Change in temperature (C) from baseline to at each follow-up assessment

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Month 1 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 2 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 3 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 4 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 5 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 6 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 7 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 8 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 9 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 10 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 11 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 12 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.9.5 Listing of vital signs

Note: Similar Tables 14.3.2.4, 14.3.2.6, 14.3.2.8 for heart rate, diastolic, and systolic blood pressure

will be produced, respectively.

# 14.3.3 Height

Table 14.3.3.1 Height (cm) at each assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Baseline | XX | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 1 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 2 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 3 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 4 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 5 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 6 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 7 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 8 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 9 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 10 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 11 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 12 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |

Table 14.3.3.2 Change in height (cm) from baseline to at each follow-up assessment

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Month 1 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 2 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 3 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 4 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 5 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 6 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 7 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 8 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 9 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 10 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 11 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 12 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |

Table 14.3.3.3 LS Means for change in height (cm) from ANCOVA model at Month 12

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | Xx | XX | |
| | LS Mean ± SE | LS Mean ± SE | LS Mean ± SE | |
| Month 12 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |

Data source: 16.2.9.5 Listing of vital signs

Table 14.3.3.4 Trend analysis for height (cm) over time

| Rate of change per month | Deferiprone | Placebo | Deferiprone<br>minus Placebo | P-value |
|---|---|---|---|---|
| Mean ± SE | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | 0.xxxx |

Data source: 16.2.9.5 Listing of vital signs

Table 14.3.3.5 Z score analysis for height (cm)

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Baseline | XX | $x.x \pm x.x (x.x, x.x)$ | xx | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |
| Month 12 | xx | $x.x \pm x.x (x.x, x.x)$ | xx | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |
| Change | XX | $x.x \pm x.x (x.x, x.x)$ | XX | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |

# 14.3.4 Weight

Table 14.3.4.1 Weight (kg) at each assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Baseline | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 1 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 2 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 3 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 4 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 5 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 6 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 7 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 8 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 9 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 10 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 11 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 12 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |

Table 14.3.4.2 Change in weight (kg) from baseline to at each follow-up assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Month 1 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 2 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 3 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 4 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 5 | xx | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 6 | xx | $xxx \pm xxx (xxx, xxx)$ | xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 7 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 8 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 9 | XX | $xxx \pm xxx (xxx, xxx)$ | XX | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 10 | xx | $xxx \pm xxx (xxx, xxx)$ | Xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 11 | XX | $xxx \pm xxx (xxx, xxx)$ | Xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |
| Month 12 | XX | $xxx \pm xxx (xxx, xxx)$ | Xx | $xxx \pm xxx (xxx, xxx)$ | 0.xxxx |

Table 14.3.4.3 LS Means for change in weight (kg) from ANCOVA model at Month 12

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | XX | XX | |
| | LS Mean ± SE | LS Mean $\pm$ SE | LS Mean ± SE | |
| Month 12 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |

Data source: 16.2.9.5 Listing of vital signs

Table 14.3.4.4 Trend analysis for weight (kg) over time

| Rate of change per month | Deferiprone | Placebo | Deferiprone<br>minus Placebo | P-value |
|---|---|---|---|---|
| Mean ± SE | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | 0.xxxx |

Data source: 16.2.9.5 Listing of vital signs

Table 14.3.4.5 Z score analysis for weight (kg)

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Baseline | XX | $x.x \pm x.x (x.x, x.x)$ | Xx | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |
| Month 12 | XX | $x.x \pm x.x (x.x, x.x)$ | Xx | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |
| Change | XX | $x.x \pm x.x (x.x, x.x)$ | Xx | $x.x \pm x.x (x.x, x.x)$ | 0.xxxx |

#### 14.3.5 Concomitant medications

Table 14.3.5.1 Concomitant medications

| | Deferiprone | Placebo | Total |
|----------------|------------------|----------------|----------------|
| | (N) | (N) | (N) |
| | | Exposure | Exposure |
| | Exposure | (Patient- | (Patient- |
| | (Patient-years): | years): | years): |
| | x.xx | X.XX | X.XX |
| | Total Patients | Total Patients | Total Patients |
| | Reporting: xx | Reporting: xx | Reporting: xx |
| Preferred Name | n Patients (%) | n Patients (%) | n Patients (%) |
| ccccc | x (x.x) | x (x.x) | x (x.x) |
| ccccc | x (x.x) | x (x.x) | x (x.x) |
| ccccc | x (x.x) | x (x.x) | x (x.x) |

Data source: 16.2.9.9 Listing of concomitant medications

## 14.3.6 Laboratory data

## 14.3.6.1 Hematology

Table 14.3.6.1.1 Hemoglobin at each assessment

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Baseline | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 1 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 2 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 3 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 4 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| | | Weekly | up to 6 | months | 1 |
| Week 28 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 30 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 32 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 36 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Biweekly until termination from the study | | | | | |

Data source: 16.2.8.1 Listing of hematology

Note: Similar tables will be produced for total WBC count, ANC, MCV, and platelet count.

Table 14.3.6.1.2 Change in hemoglobin from baseline to at each follow-up assessment

| | | Deferiprone | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Week 1 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 2 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 3 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 4 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| | | Weekly t | ip to 6 | months | |
| Week 28 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 30 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 32 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Week 36 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | Xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| | Biweekly until termination from the study | | | | |

Data source: 16.2.8.1 Listing of hematology

Note: Similar tables will be produced for total WBC count, ANC, MCV, and platelet count.

Table 14.3.6.1.3 Shift table for hemoglobin at baseline vs last assessment: deferiprone group

| | | Baseline | | | |
|---|---|---|---|---|---|
| | N (%) | Low | Normal | High | P-value (McNemar-Bowker's test) |
| Last assessment | Low | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | Normal | xx (xx) | xx (xx) | xx (xx) | |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Data source: 16.2.8.1 Listing of hematology

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

Table 14.3.6.1.4 Shift table for hemoglobin at baseline vs last assessment: placebo group

| | | Baseline | | | |
|---|---|---|---|---|---|
| | N (%) | Low | Normal | High | P-value (McNemar-Bowker's test) |
| Last assessment | Low | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | Normal | xx (xx) | xx (xx) | xx (xx) | |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Data source: 16.2.8.1 Listing of hematology

Note: Similar tables will be produced for total white blood cell (WBC), absolute neutrophil count (ANC), and platelets.

## 14.3.6.2 Biochemistry

Table 14.3.6.2.1 Albumin at each assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Baseline | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 1 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 3 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 6 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 9 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 12 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.8.4 Listing of biochemistry

Note: Similar tables will be produced for total protein, GGT, glucose, bilirubin (total, direct, and indirect), AST, ALT, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, and zinc.

Table 14.3.6.2.2 Change in albumin from baseline to at each follow-up assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (T-<br>test) |
| Month 1 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 3 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 6 | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | xx | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 9 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 12 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.8.4 Listing of biochemistry

Note: Similar tables will be produced for total protein, GGT, glucose, bilirubin (total, direct, and indirect), AST, ALT, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, and zinc.

Table 14.3.6.2.3 Shift table for albumin at baseline vs last assessment: deferiprone group

| | | Baseline | | | |
|---|---|---|---|---|---|
| | N (%) | Low | Normal | High | P-value (McNemar-Bowker's test) |
| Last assessment | Low | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | Normal | xx (xx) | xx (xx) | xx (xx) | |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Data source: 16.2.8.4 Listing of biochemistry

Note: Similar tables will be produced for total protein, GGT, glucose, bilirubin (total, direct, and indirect), AST, ALT, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, and zinc.

Table 14.3.6.2.4 Shift table for albumin at baseline vs last assessment: placebo group

| | | Baseline | | | |
|---|---|---|---|---|---|
| | N (%) | Low | Normal | High | P-value (McNemar-Bowker's test) |
| Last assessment | Low | xx (xx) | xx (xx) | xx (xx) | |
| | Normal | xx (xx) | xx (xx) | xx (xx) | 0.xxxx |
| | High | xx (xx) | xx (xx) | xx (xx) | |

Data source: 16.2.8.4 Listing of biochemistry

Note: Similar tables will be produced for total protein, GGT, glucose, bilirubin (total, direct, and indirect), AST, ALT, blood urea nitrogen, calcium, creatinine, total iron binding capacity, serum iron, and zinc.

Table 14.2.6.2.5 Percent of patients who had ALT > 2 x ULN, 3 x ULN, or 5 x ULN during the study

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|---|---|---|---|
| $ALT > 2 \times ULN$ | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| $ALT > 3 \times ULN$ | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| ALT > 5 x ULN | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

Table 14.2.6.2.6 Percent of patients who had AST > 2 x ULN, 3 x ULN, or 5 x ULN during the study

| | Deferiprone | Placebo | P-value<br>(Fisher's exact test) |
|---|---|---|---|
| $AST > 2 \times ULN$ | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| AST > 3 x ULN | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |
| AST > 5 x ULN | xx% (xx / xx) | xx% (xx / xx) | 0.xxxx |

#### 14.3.7 Prolactin

Table 14.3.7.1 Prolactin at each assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | Mean ± SD (Min, Max) | P-value (t-test) |
| Pre-dose | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Post-dose | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |
| Month 12 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.8.5 Listing of prolactin

Table 14.3.7.2 Change in prolactin from pre-dose to Month 12

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean $\pm$ SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Month 12 | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | XX | $xx.x \pm xx.x (xx.x,xx.x)$ | 0.xxxx |

Data source: 16.2.8.5 Listing of prolactin

Table 14.3.7.3 LS Means for change in prolactin from pre-dose to Month 12 from ANCOVA model

| | Deferiprone | Placebo | Deferiprone<br>Minus Placebo | 95% C.I. |
|---|---|---|---|---|
| N | XX | XX | XX | |
| | LS Mean ± SE | LS Mean ± SE | LS Mean ± SE | |
| Month 12 | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | $xxxx \pm xxxx$ | (xxxx, xxxx) |

Data source: 16.2.8.5 Listing of prolactin

# 14.4 Other analyses

Table 14.4.1 Compliance (%) at each assessment

| | Deferiprone | | | Placebo | |
|---|---|---|---|---|---|
| | N | Mean ± SD (Min, Max) | N | $Mean \pm SD (Min, Max)$ | P-value (t-test) |
| Month 1 | XX | $xx \pm xx (xx, xx)$ | XX | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 2 | XX | $xx \pm xx (xx, xx)$ | XX | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 3 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 4 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 5 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 6 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 7 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 8 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 9 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 10 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 11 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |
| Month 12 | xx | $xx \pm xx (xx, xx)$ | xx | $xx \pm xx (xx, xx)$ | 0.xxxx |

Data source: 16.2.5.1 Listing of compliance

Table 14.4.2 Overall mean of transfusional iron input (mg/kg/day) during the study

| | Deferiprone | | Placebo | | |
|---|---|---|---|---|---|
| | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value (t-test) |
| Overall mean of transfusional iron input (mg/kg/day) during the study | XX | $xx.x \pm xx.x$<br>(xx.x, xx.x) | XX | $xx.x \pm xx.x$<br>(xx.x, xx.x) | 0.xxxx |

Data source: 16.2.9.7 Listing of transfusion

Table 14.4.3 Overall mean of total daily dose (mg/kg/day) during the study

| | Deferiprone | | Placebo | | |
|---|---|---|---|---|---|
| | N | Mean ± SD<br>(Min, Max) | N | Mean ± SD<br>(Min, Max) | P-value (t-test) |
| Overall mean of total daily dose (mg/kg/day) during the study | XX | $xx.x \pm xx.x$ $(xx.x, xx.x)$ | XX | $xx.x \pm xx.x$ $(xx.x, xx.x)$ | 0.xxxx |

Data source: 16.2.9.8 Listing of exposure

Table 14.4.4 Patient exposure to study medication

| | Deferiprone | Placebo |
|------------------------------|-------------|------------|
| Total Patients Exposed [N] | XX | XX |
| Total Patient-Years Exposure | XXX | XXX |
| Length of Exposure (years) | | |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

Data source: 16.2.9.8 Listing of exposure

Table 14.4.5 Duration of study drug exposure

| | Deferiprone | Placebo |
|-----------------------------|-------------|-----------|
| Duration of Exposure [n(%)] | | |
| Any Exposure | xx (xx.x) | xx (xx.x) |
| >= 1 Month | xx (xx.x) | xx (xx.x) |
| >= 2 Months | xx (xx.x) | xx (xx.x) |
| >= 3 Months | xx (xx.x) | xx (xx.x) |
| >= 4 Months | xx (xx.x) | xx (xx.x) |
| >= 5 Months | xx (xx.x) | xx (xx.x) |
| >= 6 Months | xx (xx.x) | xx (xx.x) |
| >= 9 Months | xx (xx.x) | xx (xx.x) |
| >= 12 Months | xx (xx.x) | xx (xx.x) |

Data source: 16.2.9.8 Listing of exposure